CLINICAL TRIAL: NCT04962295
Title: China Imaging-based Biobank of Cerebral Small Vessal Diseases
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021248
Record Dates: First submitted 2021-06-27; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Small Vessel Diseases
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cerebral Small Vessel Diseases group: CSVD patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to build a national image-based comprehensive evaluation platform of CSVD through longitudinal collection of imaging based medical data of patients with cerebral small vessel diseases (CSVD). On this basis, the new classification and diagnostic criteria of CSVD are proposed, and the risk prediction model of CSVD is established. By evaluating the prognostic factors of CSVD, early identification of high-risk CSVD population.

DETAILED DESCRIPTION:
The purpose of this study is to build a national image-based CSVD comprehensive evaluation platform by collecting the medical data of patients with cerebral small vessel diseases (CSVD) based on imaging longitudinally, and to evaluate the risk factors of each type of CSVD, as well as imaging signs, cognition, gait, autonomic nervous system and hemodynamics, sleep, sleep, and so on The outcome of emotion and fundus. In the fields of imaging, molecular and neurocognitive function, we explored the etiology and pathophysiological mechanism of CSVD, proposed new classification and diagnostic criteria of CSVD, and established the risk prediction model of CSVD. By evaluating the prognostic factors of CSVD, early identification of high-risk CSVD population, in order to reduce the burden of CSVD in China in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. SVD lesions can be seen on MRI of the head

   * White matter hyperintensity, Fazekas score ≥ 2
   * Fazekas=1 has more than 2 vascular risk factors (hypertension, hyperlipidemia, diabetes, obesity, smoking, and other vascular events except stroke).
   * Fazekas = 1 and combined with lacunar focus
   * Imaging findings suggest new subcortical lacunar infarction
3. Daily life independence (MRS ≤ 2)
4. Sign informed consent

Note: the imaging definition of small vessel disease refers to the strong guideline

1. The total score of Fazekas was 6, which was the sum of Fazekas scores of subcortical and periventricular white matter lesions.
2. New subcortical lacunar infarction: head MRI examination, subcortical, basal ganglia or brain stem DWI showed high signal (ADC diffusion limited) lesions with diameter < 20 mm, with or without corresponding clinical symptoms; There were new clinical symptoms. FLAIR sequence of head MRI showed flair hyperintense lesions (diameter < 20 mm) in subcortical, basal ganglia or pons.

Exclusion Criteria:

1. In acute cerebral infarction, the lesions showed high signal intensity on DWI, and the diameter was more than 20 mm
2. Acute cerebral hemorrhage
3. Acute subarachnoid hemorrhage, or previous history of cerebrovascular malformation or aneurysmal subarachnoid hemorrhage,

   Or untreated aneurysms (> 3mm in diameter) were found
4. Neurodegenerative diseases, such as AD and PD, have been diagnosed
5. There are clear non angiogenic white matter lesions, such as multiple sclerosis, adult white matter dysplasia, metabolic encephalopathy

   Diseases, etc
6. Mental disorders diagnosed according to DSM-V diagnostic criteria
7. Contraindications of MRI examination (such as claustrophobia)
8. With severe organic diseases, such as malignant tumor, the expected survival time is less than 5 years
9. Due to geographical or other reasons can not cooperate to complete the follow-up
10. Patients also participated in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cerebral Small Vessal Diseases patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of patients with each diagnosis. | At discharge, usually within two weeks.
  Detailed diagnosis of the patient's disease.

SECONDARY OUTCOMES:
mRS score | during 5 years after diagnosis
  mRS score of patients
New adverse vascular events | during 5 years after diagnosis
  New adverse vascular events

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China